CLINICAL TRIAL: NCT04581499
Title: Applying Technology-Enabled Contingency Management for Alcohol Use Disorder at Scale
Brief Title: Tech-Enabled CM for AUD at Scale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DynamiCare Health (Industry)
Collaborators: RAND (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCH002; 2R44AA026234-02 (NIH); 5R44AA026234-03 (NIH)
Record Dates: First submitted 2020-09-15; First posted 2020-10-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence; Drug Dependence
Keywords: contingency management; motivational incentives; cognitive behavioral therapy; CBT; recovery; recovery coach; recovery coaching; telehealth; digital therapeutic; remote monitoring; drug testing; breathalyzer; Medicaid; alcoholism; alcohol abuse; addiction
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Random-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DynamiCare Motivation Support Program (Experimental): Intervention Group members will receive 32 weeks of remote Contingency Management (CM; financial motivational incentives), Recovery Coaching, substance testing, appointment reminding/tracking, and in-app Cognitive Behavioral Therapy (CBT). After 32 weeks, coaching, testing, appointment tracking and CBT will continue until an overall 12 months in the project is completed.
  Interventions: Combination Product: DynamiCare Motivation Support Program
- Untreated or Routine Care Control Group (Other): Control participants will receive substance tests at the same frequency as Intervention participants, and the same incentive amounts for tests as treatment participants. Controls' payments, however, will not be contingent on positive/negative results, but rather only on valid, on-time submission. Controls will not receive coaching, CBT or rewards for appointments.
  Interventions: Other: Untreated or Routine Care Control Group

INTERVENTIONS:
Combination Product: DynamiCare Motivation Support Program — DynamiCare is an evidence-based, multi-service platform that combines software, smartphone and pocket-sized alcohol and drug testing hardware, and recovery services, designed to remotely deliver evidence-based methodologies to facilitate people's motivation and accountability to overcome alcohol, nicotine and other drug use disorders, whether in formal treatment or not.
  Arms: DynamiCare Motivation Support Program
Other: Untreated or Routine Care Control Group — No specific intervention, i.e., research participation plus any community-based treatment the individual seeks to obtain.
  Arms: Untreated or Routine Care Control Group

SUMMARY:
This Phase II Small Business Innovative Research (SBIR) project is a clinical effectiveness and cost-effectiveness random controlled trial (RCT) of DynamiCare Health's innovative smartphone/smart debit card remote digital coaching program, which integrates Contingency Management, Recovery Coaching, and cognitive behavioral therapy (CBT), to address alcohol use disorder (AUD) in 300 adults.

DETAILED DESCRIPTION:
This application proposes to continue clinical effectiveness and cost-effectiveness testing of the DynamiCare Health platform. This is an innovative smartphone-based digital coaching program that offers remotely-delivered contingency management (CM), Recovery Coaching, and cognitive behavioral therapy (CBT) content to address alcohol use disorder (AUD). CM, which uses financial incentives to reward abstinence and treatment attendance, is one of the most effective, evidence-based, and overlooked intervention for substance use disorders (SUD). DynamiCare, through its remote delivery system, has addressed the logistical barriers to adoption, and now seeks, through this proposal, to drive payer adoption. Our Phase 1 preliminary data shows that the intervention is acceptable and can be highly effective when delivered as a supplemental therapy to persons with AUD enrolled in treatment. Phase 2 proposes to partner with Medicaid to deploy and test the fully developed intervention in an RCT among individuals with AUD (n=300). Our goals are to: 1) Deploy the DynamiCare CM and digital coaching program at scale among Medicaid members with AUD; 2) determine clinical effectiveness; and 3) evaluate the cost-effectiveness and return-on-investment from the payer perspective. This study design addresses a lack in the CM literature of empirical evidence on the cost-savings for payers from CM. If CM can be shown to create cost-savings for payers, the final barrier to widespread adoption would fall. Overall, this Phase 2 project, which follows a highly successful Phase 1, will provide critical data to advance the utility of this innovative digital platform as it is deployed in the real world to help the millions of people with AUD.

ELIGIBILITY:
Inclusion Criteria:

Participants in the study must have Alcohol Use Disorder (AUD) and:

1. Be >18 years old
2. Meet the DSM-5 criteria for current (past year) AUD, or be recommended for care in the ASAM CO-Triage assessment
3. Have consumed at least one alcoholic beverage within the last 10 days, according to self-report
4. Speak English
5. Have an Android or iOS smartphone.

Exclusion Criteria:

1. Participants with current suicidal intent will be excluded as they require a higher level of care that cannot be provided by DynamiCare and our Recovery Coaches (hence, these individuals will be directly referred for clinical evaluation).
2. Participants with ASAM CO-Triage level needs higher than Level 3.1 (e.g., greater than community-based, working halfway house) and not receiving addiction treatment will be excluded because they require inpatient treatment. Once the participant has received treatment, Recovery Coaches will reach out again to re-enroll the participant in the study if the participant wishes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are eligible
Enrollment: 236 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Alcohol Use | 32 weeks
  The primary outcome measure is alcohol use, in terms of the number of weeks of abstinence confirmed by DynamiCare Breathalyzer tests and self-report.

SECONDARY OUTCOMES:
Engagement | 32 weeks
  Percent of available funds earned as a composite measure.
Retention | 32 weeks
  Monthly rates of retention in the program.
Drug Use Clinical Effectiveness | 32 weeks
  Measured by DynamiCare saliva drug test results and weekly self-report.
Cost-effectiveness | 12 months
  Medicaid healthcare utilization claims costs vs. prior 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Eric E Gastfriend, MBA, Principal Investigator — DynamiCare Health Inc.
Locations (1):
- DynamiCare Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Press release describing study launch and Vermont Medicaid's Chief Medical Officer's rationale. — https://www.prnewswire.com/news-releases/vt-medicaid-gets-creative-on-addiction-during-covid-19-301108477.html